CLINICAL TRIAL: NCT04111263
Title: Efficacy of a Gut-microbiota Targeted Nutritional Intervention for Promoting Gut Barrier Integrity During Short-term Exposure to Hypobaric Hypoxia.
Brief Title: Gut-microbiota Targeted Nutritional Intervention for Gut Barrier Integrity at High Altitude
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Army Research Institute of Environmental Medicine (U.S. Federal Agency)
Collaborators: US Army Combat Capabilities Development Command- Soldier Center (Unknown); Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency); University of Reading (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 19-02-HC; M-10783 (Other: USMRMC)
Record Dates: First submitted 2019-07-02; First posted 2019-10-01 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Gastrointestinal Injury; Acute Mountain Sickness
Keywords: Microbiome; Intestinal permeability; Cognition; Immune; Fiber; Military; Altitude; Polyphenol
MeSH Terms: conditions — Altitude Sickness | interventions — Sea Level Rise

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- PL+SHAM (Sham Comparator): Placebo intervention + sea level exposure
  Interventions: Dietary Supplement: Placebo; Other: Sea level
- PL+HA (Placebo Comparator): Placebo intervention + high altitude exposure
  Interventions: Dietary Supplement: Placebo; Other: High altitude
- FP+HA (Experimental): Fiber and polyphenol supplementation + high altitude exposure
  Interventions: Dietary Supplement: FP; Other: High altitude

INTERVENTIONS:
Dietary Supplement: FP — Fiber and polyphenol blend
  Arms: FP+HA
Dietary Supplement: Placebo — Matched placebo
  Arms: PL+HA; PL+SHAM
Other: High altitude — Simulated high altitude in altitude chamber using hypobaric hypoxia
  Arms: FP+HA; PL+HA
Other: Sea level — Sea level environment in altitude chamber
  Arms: PL+SHAM

SUMMARY:
The aim of this randomized, crossover clinical trial is to determine the efficacy of a gut microbiota-targeted nutritional intervention containing a blend of fermentable fibers and polyphenols (FP) for mitigating increases in GI permeability, and decrements in immune function and neuropsychologic performance following rapid ascent to simulated high altitude. Fifteen healthy young adults will participate in each of three study phases that include a 14-day supplementation period in which participants will consume 1 of 2 supplement bars: placebo (PL, will be consumed during 2 phases) and FP supplementation (will be consumed during one phase only). During the final 2-d of each phase, participants will live in a hypobaric chamber under sea level or high altitude conditions.

DETAILED DESCRIPTION:
The collection of microbes inhabiting the human gastrointestinal (GI) tract, known as the gut microbiota, is increasingly recognized as a mediator of GI, immunologic, and neuropsychologic responses to various environmental and physiologic stressors. The hypobaric hypoxia characteristic of high altitude environments is a stressor that has recently been associated with increased GI permeability, and which has been shown to cause decrements in immune, neuropsychological and physical function. To what extent modulation of the human gut microbiota can mitigate these responses during high altitude exposure is undetermined. The aim of this randomized, crossover clinical trial is to determine the efficacy of a gut microbiota-targeted nutritional intervention containing a blend of fermentable fibers and polyphenols (FP) for mitigating increases in GI permeability, and decrements in immune function and neuropsychologic performance following rapid ascent to simulated high altitude. Fifteen healthy young adults will participate in each of three study phases in random order. Each phase will include a 14-day supplementation period in which participants will consume 1 of 2 supplement bars: placebo (PL, will be consumed during 2 phases) and FP supplementation (will be consumed during one phase only). During the final 2-d of each phase, participants will live in a hypobaric chamber. During one phase the chamber environment will mimic low-altitude conditions (SHAM). During two phases the chamber environment will mimic the barometric pressure at Pike's Peak CO (460 mmHg; HA).

ELIGIBILITY:
Inclusion criteria:

* Men and women aged 18 - 39 years (active duty personnel who are 17 yr of age will also be allowed to participate)
* In good health
* Physically active
* For active duty, passed most recent body composition assessment; for civilians, body mass index (BMI) ≤ 30.0 kg/m2.
* Self-reports having a bowel movement at least as frequently as every-other-day
* Self-reports normal vision (with or without glasses) and hearing

Exclusion Criteria:

* Born at altitudes greater than 2,100 m (~7,000 feet)
* Living in areas that are more than 1,200 m (~4,000 feet), or have traveled to areas that are more than 1,200 m for five days or more within the last 2 mo
* Pregnant, expecting to become pregnant during study, or breastfeeding
* Any of the following medical conditions:

  1. Musculoskeletal injuries that compromise exercise capability
  2. Metabolic or cardiovascular abnormalities (e.g., kidney disease, diabetes, cardiovascular disease, etc.)
  3. Suspected or known strictures, fistulas, or physiological/mechanical GI obstruction
  4. Evidence of apnea or other sleeping disorders
  5. Evidence of prior high altitude pulmonary or cerebral edema diagnosis
  6. Disease of the GI tract including, but not limited to diverticulitis, inflammatory bowel disease, peptic ulcer disease, Crohn's disease, ulcerative colitis
  7. Anemia or Sickle Cell Anemia/Trait
  8. Alcoholism or other substance abuse issues
  9. History of gastric bezoar
  10. Swallowing disorders; severe dysphagia to food or pills
  11. Implanted or portable electro-mechanical medical devices
  12. Allergy to skin adhesive
* Past GI surgery
* Colonoscopy within 3 months of study participation
* Taking prescription medications other than a contraceptive (unless approved by Medical Office and study PI)
* Regular use of over-the-counter medications (including antacids, laxatives, stool softeners, and anti-diarrheals) unless approved by Medical Office and study PI
* Any use of antibiotics, except topical antibiotics, within 3 months of study participation
* Not willing to refrain from using non-steroidal anti-inflammatory medications (NSAIDs) or antihistamine during the study
* Not willing to stop consumption of prebiotic- or probiotic-containing supplements (e.g.,VSL#3, PRO-15, etc.), or other dietary supplements at least 2 weeks before and throughout study participation
* Not willing to stop consumption of probiotic-containing foods (e.g., yogurt, etc.) during study participation.
* Not willing to refrain from smoking any nicotine product (includes e-cigarettes), vaping, and chewing tobacco during controlled-diet periods.
* Not willing to abstain from caffeine and alcohol during controlled-diet periods.
* Allergies, intolerances, unwillingness or inability to eat provided foods and beverages
* Following vegetarian/vegan diet
* Unable to regularly sleep for 7-10 hr/night
* Any previous blood donation, within 8 weeks of the first blood draw of the study, of a volume that when combined with the amount of blood to be collected during the study would exceed 550 mL

Ages: 17 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 33 (Actual)
Dates: Start 2019-10-06 (Actual); Primary Completion 2022-11-05 (Actual); Study Completion 2022-11-05 (Actual)

PRIMARY OUTCOMES:
Difference in intestinal permeability | Study days 20, 40 and 60
  Intestinal permeability measured by the ratio of the urinary excretion of sucralose and erythrirol

SECONDARY OUTCOMES:
Difference in lipopolysaccharide binding protein concentrations | Study days 20, 21, 41, 42, 62, 63
  Fasting serum lipopolysaccharide binding protein concentration
Difference in zonulin concentrations | Study days 20, 21, 41, 42, 62, 63
  Fasting serum zonulin concentration
Difference in glucagon-like peptide-2 concentrations | Study days 20, 21, 41, 42, 62, 63
  Fasting serum glucagon-like peptide-2 concentration
Difference in intestinal fatty acid binding protein concentrations | Study days 20, 21, 41, 42, 62, 63
  Fasting and post-exercise serum intestinal fatty acid binding protein concentration
Difference in claudin-3 concentrations | Study days 20, 21, 41, 42, 62, 63
  Fasting and post-exercise serum claudin-3 concentration
Difference in S100B concentrations | Study days 20, 21, 41, 42, 62, 63
  Fasting and post-exercise serum S100B concentration
Difference in systemic inflammation | Study days 20, 21, 41, 42, 62, 63
  Fasting serum interleukin (IL) IL-6, IL-8, IL-10, IL-17, IL-1β, IL-1ra, tumor necrosis factor-α, interferon-γ concentrations
Difference in intestinal inflammation | Study days 6, 18, 21, 23, 27, 39, 42, 44, 48, 60, 63, 65
  Fecal calprotectin concentration
Difference in glucose concentrations | Study days 20, 21, 41, 42, 62, 63
  Fasting and post-exercise serum glucose concentrations
Difference in insulin concentrations | Study days 20, 21, 41, 42, 62, 63
  Fasting and post-exercise serum insulin concentrations
Difference in lactate concentrations | Study days 20, 21, 41, 42, 62, 63
  Fasting and post-exercise serum lactate concentrations
Difference in glycerol concentrations | Study days 20, 21, 41, 42, 62, 63
  Fasting and post-exercise serum glycerol concentrations
Difference in cortisol concentrations | Study days 20, 21, 41, 42, 62, 63
  Fasting and post-exercise serum cortisol concentrations
Difference in bone specific alkaline phosphatase concentrations | Study days 20, 41, 62
  Fasting serum bone specific alkaline phosphatase concentration
Difference in carboxy-terminal collagen crosslinks concentrations | Study days 20, 41, 62
  Fasting serum carboxy-terminal collagen crosslinks concentration
Difference in tartrate resistant acid phosphatase concentrations | Study days 20, 41, 62
  Fasting serum tartrate resistant acid phosphatase concentration
Difference in procollagen type 1 N-terminal propeptide concentrations | Study days 20, 41, 62
  Fasting serum procollagen type 1 N-terminal propeptide concentration
Difference in osteocalcin concentrations | Study days 20, 41, 62
  Fasting serum osteocalcin concentration
Difference in secretory immunoglobulin A concentrations | Study days 20, 21, 41, 42, 62, 63
  Secretory immunoglobulin A concentrations in tear fluid and saliva
Difference in immune cell phenotypes | Study days 21, 42, 63
  Immune cell phenotype by flow cytometry
Difference in T-cell simulated cytokine production | Study days 21, 42, 63
  T-cell simulated cytokine production by cell culture and flow cytometry
Difference in natural killer-cell cytotoxicity | Study days 21, 42, 63
  Natural killer-cell cytotoxicity by cell culture and flow cytometry
Difference in development of acute mountain sickness | Study days 20, 21, 41, 42, 62, 63
  Environmental Symptoms Questionnaire-short form. Acute Mountain Sickness will be measured multiple times daily using the Lake Louise scoring system wherein higher scores indicate more severe symptoms. AMS severity cutoffs will use mild (0.7-1.53), moderate (1.53-2.63), severe >=2.63
Difference in gastrointestinal symptoms; quality of life | Study weeks 0, 1, 2, 3, 4, 5, 6, 7, 8, 9
  Gastrointestinal symptoms measure by modified version of the gastrointestinal quality of life index wherein lower scores indicate more severe symptoms.
Difference in gastrointestinal symptoms; irritable bowel syndrome | Study weeks 0, 1, 2, 3, 4, 5, 6, 7, 8, 9
  Gastrointestinal symptoms measure by modified version of the irritable bowel syndrome symptom severity scale score wherein higher scores indicate more severe symptoms. Scored on scale of 0-500; symptom severity scored as mild (75-174), moderate (175-300), severe (>300).
Difference in appetite | Study weeks 0, 1, 2, 3, 4, 5, 6, 7, 8, 9
  Hunger, fullness, desire to eat, and prospective consumption measured by 100 mm visual analog scale. Scored from 0-100 with higher scores indicating greater sensation.
Difference in changes in mood state | Study days 20, 21, 41, 42, 62, 63
  Measured by Profile of Mood States Questionnaire; a 65-item inventory of self-reported mood states which factor into six mood sub-scales (tension/anxiety (0-36), depression/dejection (0-60), anger/hostility (0-48), vigor/activity (0-32), fatigue/inertia (0-28), confusion/bewilderment (0-28), and total mood disturbance (0-200) wherein higher scores indicate greater mood state.
Difference in changes in feeling | Study days 20, 21, 41, 42, 62, 63
  Measured by Feeling Scale; a one-item inventory measuring the extent to which participants feel pleasant or unpleasant. Higher scores indicate more unpleasant feeling. Scored from -5 (very bad) to 5 (very good)
Difference in changes arousal | Study days 20, 21, 41, 42, 62, 63
  Measured by Felt Arousal Scale; a one-item inventory measuring the extent to which participants feel aroused. Higher scores indicate greater arousal (low=1 to high =6).
Difference in willingness to take risks | Study days 20, 21, 41, 42, 62, 63
  Measured by Evaluation of Risks Questionnaire; a 24-item questionnaire providing scores on five scales: self-control, danger seeking, energy, impulsivity, and invincibility.
Difference in risk taking behavior | Study days 7, 20, 21, 41, 42, 62, 63
  Measured by Balloon Analogue Risk Task
Difference in resting metabolic rate | Study days 7, 21, 42, 63
  Resting metabolic rate measured by indirect calorimetry
Difference in physical activity energy expenditure | Study days 20, 21, 41, 42, 62, 63
  Energy expenditure measured by indirect calorimetry during 60-minute steady state exercise
Difference in gastrointestinal transit time | Study days 20, 41, 62
  Gastric, small intestine and large intestine transit time measured by SmartPill
Difference in gastrointestinal pH | Study days 20, 41, 62
  Gastric, small intestine and large intestine pH measured by SmartPill
Difference in changes in working memory | Study days 20, 21, 41, 42, 62, 63
  Measured by N-Back task before, during and after exercise
Difference in changes in spatial working memory | Study days 20, 21, 41, 42, 62, 63
  Measured by emotional Interference task before, during and after exercise
Difference in changes in spatial memory | Study days 20, 21, 41, 42, 62, 63
  Measured by Matching to Sample test in the morning and afternoon
Difference in change in reaction time | Study days 20, 21, 41, 42, 62, 63
  Measured by reaction time task before, during and after exercise
Difference in change in response inhibition | Study days 20, 21, 41, 42, 62, 63
  Measured by Go/No-Go task before, during and after exercise
Difference in vigilance | Study days 20, 21, 23, 41, 42, 44, 62, 63, 65
  Measured by scanning visual vigilance task
Difference in simple visual reaction time | Study days 20, 21, 23, 41, 42, 44, 62, 63, 65
  Measured by psychomotor vigilance test
Difference in language-based logical reasoning | Study days 20, 21, 23, 41, 42, 44, 62, 63, 65
  Measured by grammatical Reasoning task
Difference in ambulatory vigilance | 48-hours/day during study weeks 0, 2, 3, 5, 6, 8, 9
  Measured by wrist-worn vigilance monitor
Difference in fecal short chain fatty acids | Study days 6, 18, 21, 23, 27, 39, 42, 44, 48, 60, 63, 65
  Fecal short chain fatty acid concentrations
Difference in gut microbiota composition | Study days 6, 18, 21, 23, 27, 39, 42, 44, 48, 60, 63, 65
  Fecal bacterial community diversity and relative abundance measured by 16S rRNA gene sequencing
Differences in microRNA concentrations | Study days 20, 21, 41, 42, 62, 63
  Fasting and post-exercise circulating and exosomal microRNA

CONTACTS AND LOCATIONS:
Overall Officials: J. Philip Karl, PhD, Principal Investigator — United States Army Research Institute of Environmental Medicine
Locations (1):
- USARIEM, Natick, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2022-06-28): https://cdn.clinicaltrials.gov/large-docs/63/NCT04111263/ICF_000.pdf